CLINICAL TRIAL: NCT00428922
Title: Phase II Trial of Trastuzumab (Herceptin), Bevacizumab, and Docetaxel (Taxotere) Trial in Stage IV Metastatic Breast Cancer (MBC) Patients
Brief Title: Trastuzumab (Herceptin), Bevacizumab, and Docetaxel (Taxotere) Trial in Stage IV Metastatic Breast Cancer (MBC) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bhuvaneswari Ramaswamy (Other)
Collaborators: Genentech, Inc. (Industry); Case Comprehensive Cancer Center (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Bhuvaneswari Ramaswamy, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-06027; NCI-2011-03219 (Registry Identifier: Clinical Trial Reporting Program (CTRP))
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer
Keywords: Metastatic; Breast Cancer; MBC
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Trastuzumab; Bevacizumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Trastuzumab, Bevacizumab, and Docetaxel (Experimental): Trastuzumab [6mg/kg], Bevacizumab [15mg/kg], and Docetaxel [75 mg/M²]
  Interventions: Drug: Trastuzumab; Drug: Bevacizumab; Drug: Docetaxel

INTERVENTIONS:
Drug: Trastuzumab — administered every three weeks on day 1, every 21 days. The dose given will be 6 mg/kg. The initial loading dose is 8mg/kg and is administered as a 90-minute infusion. Thereafter, the maintenance dose is 6mg/kg every three weeks administered as a 30 minute infusion (unless the treating physician indicates a longer infusion duration is warranted). Trastuzumab is given prior to bevacizumab. Trastuzumab is to be continued until disease progression or unacceptable toxicity.
  Other Names: Herceptin
Drug: Bevacizumab — administered every three weeks on day 1, every 21 days. The dose given will be 15 mg/kg. The initial dose is administered over 90 minutes. If the first infusion is well tolerated, the second dose is given over 60 minutes, and if that is well tolerated, then subsequent doses may be given over 30 minutes. Avastin is given after trastuzumab and prior to docetaxel.
  Other Names: Avastin
Drug: Docetaxel — administered every three weeks on day 1, every 21 days. The dose given will be 75 mg/M². All doses of docetaxel are administered over 60 minutes. Docetaxel is given after trastuzumab and bevacizumab.
  Other Names: Taxotere

SUMMARY:
The primary objectives are to determine the progression-free survival (PFS) and to evaluate safety of the trastuzumab, bevacizumab and docetaxel regimen.

DETAILED DESCRIPTION:
Rationale: Antibodies are proteins that are normally part of the immune system that bind to foreign agents in the body. Researchers manufacture antibodies outside of the human body that bind to specific targets such as proteins in cancer cells. Herceptin is a monoclonal antibody that binds to the human epidermal growth factor receptor (HER-2), and can kill HER2-positive cancer cells. Herceptin is used to treat breast cancer that is HER2-positive, and has spread after treatment with other drugs. Bevacizumab is a signal transduction inhibitor that works by preventing the growth of new blood vessels from surrounding tissue into tumors. Bevacizumab specifically inhibits the vascular endothelial growth factor (VEGF), a substance made by cells that stimulates new blood vessel formation. Research indicates that HER-2 signaling helps to induce VEGF expression. Therefore, cancer treatments targeting both HER-2 and VEGF may improve anti-cancer efficacy in patients. Docetaxel is a chemotherapy agent used against breast and other types of cancer. The current study builds on previous research suggesting the safety and potential for efficacy with combination trastuzumab, bevacizumab, and docetaxel.

Purpose: The primary objectives are to determine the progression free survival and evaluate the safety of trastuzumab, bevacizumab, and docetaxel. Secondary objectives are to assess early changes in circulating tumor cells and circulating endothelial cells as predictors of progression free survival and clinical benefit, as well as to determine the overall clinical benefit rate.

Treatment: Study participants will be given trastuzumab, bevacizumab, and docetaxel. All study drugs will be given through intravenous infusions once every 21 days. A cycle is considered 3 weeks. A minimum of 6 study treatment cycles is required unless study participants experience disease growth or intolerable toxicity. The decision to stop docetaxel after 6 cycles is up to the discretion of the treating physician and the patient. Study participants who are deriving a benefit from the study drugs may continue on trastuzumab and bevacizumab alone. Several tests and exams will be given throughout the study to closely monitor study participants.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer with evidence of metastatic disease
* HER2 3+ or FISH (fluorescent in situ hybridization)+
* Age ≥ 18 years
* No prior trastuzumab, except as given in the adjuvant or neoadjuvant setting.
* No prior chemotherapy in the metastatic setting.

Exclusion Criteria:

* CNS (central nervous system) metastases
* Prior radiation therapy within the last 4 weeks
* Pregnant (positive pregnancy test) or lactating women
* Major surgical procedure, open biopsy, non-healing wounds, or significant traumatic injury within 28 days prior to starting study or anticipation of need for major surgical procedure during the study
* Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to start of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-06-14 (Actual); Primary Completion 2012-11-01 (Actual); Study Completion 2017-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhuvaneswari Ramaswamy, MD, Principal Investigator — Ohio State University
Locations (3):
- United States (3):
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Puhalla S, Mrozek E, Young D, Ottman S, McVey A, Kendra K, Merriman NJ, Knapp M, Patel T, Thompson ME, Maher JF, Moore TD, Shapiro CL. Randomized phase II adjuvant trial of dose-dense docetaxel before or after doxorubicin plus cyclophosphamide in axillary node-positive breast cancer. J Clin Oncol. 2008 Apr 1;26(10):1691-7. doi: 10.1200/JCO.2007.14.3941. Epub 2008 Mar 3. PMID 18316792
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: September 2007 and November 2012
Period: Overall Study
Arm/Group | Trastuzumab, Bevacizumab, and Docetaxel
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Trastuzumab, Bevacizumab, and Docetaxel
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 54 [38 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 0
Region of Enrollment [Number; unit: patients]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) and to Evaluate Safety of the Trastuzumab, Bevacizumab and Docetaxel Regimen.
Description: The trial was designed as a single-stage phase II rather then usual two-stage design because of the progression free survival (PFS) primary endpoint, as it is impractical to wait to assess PFS for patients in the first stage. We will consider a PFS of 50% at twelve months (median PFS of 12 months) or less uninteresting and a PFS of 70% at twelve months (median PFS of twenty months) worthy of pursuing the regimen in a future trials. The single-stage design is as follows: p0=0.50, p1=0.70, α=0.10, β= 0.10. This leads to a total sample size of 39 patients, 24 or higher of who are progression-free at 12 months.
Time Frame: up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab, Bevacizumab, and Docetaxel
Number analyzed (Participants) | 26
months | 14.3 [9.3 to 35]

2. Secondary Outcome: Changes in CTCs as Predictors of PFS and Clinical Benefit
Description: Circulating tumor cells (CTCs) evaluated at baseline (day 1 of treatment) and after 1 treatment cycle (day 22 prior to cycle 2 treatment).
Time Frame: Day 1 and Day 22
Population: Due to sample size, could not perform any statistical analysis to correlate the baseline CTCs with PFS and response rate. Samples only available for 50% of the patients.
Measure: Number; unit: patients with detected CTCs
Arm/Group | Trastuzumab, Bevacizumab, and Docetaxel
Number analyzed (Participants) | 13
patients with detected CTCs | 7

3. Secondary Outcome: Overall Clinical Benefit Rate (CR+PR+SD)
Description: Defined as best response of CR or PR or stable disease for at least 24 weeks. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI and/or CT: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for a Partial Response nor sufficient increase to qualify for Progression of Disease (POD); POD, 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Complete Response (CR), Disappearance of all target lesions
Time Frame: at least 24 weeks
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Trastuzumab, Bevacizumab, and Docetaxel
Number analyzed (Participants) | 26
percent of patients | 69 [48 to 86]

4. Secondary Outcome: Changes in CECs as Predictors of PFS and Clinical Benefit
Description: Circulating endothelial cells (CECs) are to be collected day 1 prior to treatment and day 22 prior to treatment. These samples are to be collected at the PI's discretion based upon the availability of the cell processing laboratory, the patients will be informed when consented if the samples will collected or not.
Time Frame: Day 1 and Day 22
Population: CEC data was not collected and available for analysis
Arm/Group | Trastuzumab, Bevacizumab, and Docetaxel
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: NCI Common Toxicity Criteria (CTC) version 3.0 was utilize the CTC for adverse event reporting.
Arm/Group | Trastuzumab, Bevacizumab, and Docetaxel
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 26/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab, Bevacizumab, and Docetaxel (N=26)
Anemia (Blood and lymphatic system disorders) | 11 (11)
Neutropenia (General disorders) | 4 (4)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Fever without neutropenia (General disorders) | 8 (8)
Infection (Infections and infestations) | 24 (24)
Fatigue (General disorders) | 24 (24)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (21)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (19)
Abdominal Pain (Gastrointestinal disorders) | 12 (12)
Constipation (Gastrointestinal disorders) | 12 (12)
Diarrhea (Gastrointestinal disorders) | 19 (19)
Nausea (Gastrointestinal disorders) | 18 (18)
Vomiting (Gastrointestinal disorders) | 14 (14)
Rash (Skin and subcutaneous tissue disorders) | 11 (11)
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 9 (9)
decreased LVEF (Cardiac disorders) | 3 (3)
Hypertension (Vascular disorders) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16 (16)
Headaches (Nervous system disorders) | 15 (15)
Vision changes (Eye disorders) | 12 (12)
Proteinuria (Renal and urinary disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 (22)
Wound Complication (Skin and subcutaneous tissue disorders) | 2 (2)
Mucositis (Gastrointestinal disorders) | 19 (19)
Increased lacrimation (Eye disorders) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes